CLINICAL TRIAL: NCT00893594
Title: A Parallel Two Arm, Double Blinded Placebo Study, Examining the Efficacy of Sumatriptan With Naprosyn in the Treatment of Migraine With Aura
Brief Title: Efficacy of Sumatriptan With Naprosyn in Migraine With Aura
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dent Neurologic Institute (Other)
Responsible Party: Principal Investigator, Mary Kay Betz, MS RPA-C, Physician Assistant, Dent Neurologic Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 113010
Record Dates: First submitted 2009-05-04; First posted 2009-05-06 (Estimated); Last update posted 2015-02-19 (Estimated); Status verified 2015-02

CONDITIONS: Migraine With Aura
Keywords: migraine; migraine with aura; headache
MeSH Terms: conditions — Migraine with Aura; Migraine Disorders; Headache | interventions — Sumatriptan; Naproxen; sumatriptan-naproxen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): Placebo taken at onset of aura associated with migraine.
  Interventions: Drug: placebo
- 2 (Active Comparator): Sumatriptan with naprosyn taken at onset of aura associated with migraine.
  Interventions: Drug: sumatriptan with naprosyn

INTERVENTIONS:
Drug: sumatriptan with naprosyn — Subjects will be randomized before treatment. Subjects will take one sumatriptan 85mg/naprosyn 500mg tablets (Treximet) or placebo at onset of a migraine aura. Dose to be repeated at 2 hours if no effect in preventing onset of migraine pain.
  Other Names: Treximet
  Arms: 2
Drug: placebo — Subjects will be randomized before treatment. Subjects will take one sumatriptan 85mg/naprosyn 500mg tablets (Treximet) or placebo at onset of a migraine aura. Dose to be repeated at 2 hours if no effect in preventing onset of migraine pain.
  Arms: 1

SUMMARY:
This is a double-blinded placebo study, examining the efficacy of Sumatriptan with Naprosyn in the treatment of migraine with aura.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 18 to 50 years of age, inclusive.
* Patients will meet the International Headache Society (IHS) classification criteria for migraine with aura.
* Subjects must carry the diagnosis of 1-2 migraine with aura per month for at least three months before study inclusion. and migraine with aura were included in the study
* Subjects must have an onset of a visual aura that occurs 15-30 minutes before a migraine headache.
* Subjects must be able to understand and complete a migraine diary.
* Subjects must be able to distinguish a migraine with aura from other types of headache.
* Subjects must be in generally good health as confirmed by medical and medication history, baseline physical and neurological exam and vital signs.
* Female subjects must be either a) postmenopausal for one year, b)surgically sterile, c) practicing acceptable birth control for at least one month prior to screening and throughout study, or d) practicing abstinence and agree to continue same throughout study.

Exclusion Criteria:

* Subjects who have a significant systemic disease other than migraine that is equally painful or more painful.
* Subjects who have other progressive neurological disorders.
* Subjects who have more than 8 migraines or 15 headache days per month.
* Subjects who have previously taken Treximet and failed due to lack of efficacy or adverse side effects.
* Subjects who carry the diagnosis of chronic tension type headache or cluster headache based on the International Headache Society criteria.
* Subject should not have received any other investigative drug within 3 months prior to enrollment in the study.
* Subject who have the diagnosis of seizure disorder, chronic daily headache, uncontrolled hypertension, cardiovascular disease, history of stroke, basilar or hemiplegic migraine, hepatic disease, or active peptic ulcer disease.
* Subjects currently taking or in 3 months prior to study, use of prophylactic migraine medications.
* Subjects who have a known allergy to Sumatriptan or Naprosyn.
* Subjects who in the opinion of Dr. Mechtler have a condition for which they should not be enrolled in the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-10; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Primary outcome measure will be comparative percentage of patients pain free at 2 and 4 hours from initiating treatment with placebo vs treatment with Treximet (sumatriptan with naprosyn). | 2 and 4 hours

SECONDARY OUTCOMES:
Secondary outcomes will be percentage of patients with pain relief at 2 and 4 hours. | 2 and 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Laszlo L Mechtler, MD, Principal Investigator — Dent Neurologic Institute
Locations (1):
- Dent Neurologic Institute, Amherst, New York, United States